CLINICAL TRIAL: NCT02703831
Title: Single Versus Dual Spine Attending Surgeons in Complex Adult Deformity Surgery: A Cost-effectiveness Study Using Activity-based Costing
Brief Title: Single Versus Dual Spine Attending Surgeons in Complex Adult Deformity Surgery:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Norton Leatherman Spine Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-N0036
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Scoliosis, Unspecified
Keywords: adult spine deformity; time-driven activity-based costing; three-column posterior osteotomy
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual attending (Active Comparator): Two attending spine surgeons during the critical portions of the surgery
  Interventions: Procedure: Dual attending
- Single attending (Placebo Comparator): One spine attending and an assistant during the critical portions of the surgery, The assistant can be a spine fellow, a resident or a physician's assistant.
  Interventions: Procedure: Single Attending

INTERVENTIONS:
Procedure: Dual attending — Two attending spine surgeons perform surgery
  Arms: Dual attending
Procedure: Single Attending — One spine attending and an assistant perform surgery. The assistant can be a spine fellow, a resident or a physician's assistant.
  Arms: Single attending

SUMMARY:
Two recent studies showed that having two attending spine surgeons performing complex adult spine deformity surgery instead of one, decreased complications, unplanned surgeries within 30-days [Ames], 90-day readmissions, wound infection, pulmonary embolism/deep vein thrombosis and post-operative neurologic complications [Sethi]. However, both studies were retrospective and did not evaluate any cost-savings associated with having two spine surgeons instead of one performing complex spine deformity surgery.

Most cost-effectiveness studies have used traditional accounting (TA) methods to determine costs. A few cost-effectiveness studies have used time-driven activity-based costing (TDABC) [Kaplan] in medicine [Au, Balakrishnan] and none in spine surgery.

Objectives: The objectives of the study are (1) to determine if dual spine attendings reduce downstream costs compared to a single spine attending for complex spine surgeries using traditional accounting methods; and (2) to demonstrate an application of the TDABC method to evaluate the operating room phase during complex adult spinal deformity surgery and compare it to traditional accounting methods (TA).

DETAILED DESCRIPTION:
Two recent studies showed that having two attending spine surgeons performing complex adult spine deformity surgery instead of one, decreased complications, unplanned surgeries within 30-days [Ames], 90-day readmissions, wound infection, pulmonary embolism/deep vein thrombosis and post-operative neurologic complications [Sethi]. However, both studies were retrospective and did not evaluate any cost-savings associated with having two spine surgeons instead of one performing complex spine deformity surgery. With increasing scrutiny on the efficient use of health care dollars, it would be important to determine if there are any downstream cost savings to justify paying the surgeon fees of two spine attendings for these complex and high cost cases.

Most cost-effectiveness studies have used traditional accounting (TA) methods to determine costs. TA uses allocated expenses from the general ledger and payroll activity codes. These codes are derived from billable items and procedures entered into accounting software. Costs of services are grouped by cost types, across units of service.

A few cost-effectiveness studies have used time-driven activity-based costing (TDABC) [Kaplan] in medicine [Au, Balakrishnan] and none in spine surgery. TDABC allows for detailed identification of costs during all phases of a patient's care cycle. While TDABC has been used in other industries, its use has been described only a few times in health care and rarely in the operative setting [Balakrishnan]. This may be due to the large amount of manpower necessary to collect TDABC data.

Objectives: The objectives of the study are (1) to determine if dual spine attendings reduce downstream costs compared to a single spine attending for complex spine surgeries using traditional accounting methods; and (2) to demonstrate an application of the TDABC method to evaluate the operating room phase during complex adult spinal deformity surgery and compare it to traditional accounting methods (TA).

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for a complex spine adult deformity surgery.

   1. instrumented posterior fusion from the thoracic spine into the pelvis, S1 or iliac wings;
   2. and/or any three-column posterior osteotomy, either a pedicle subtraction osteotomy or a vertebral column resection.
2. Is at least 25 years of age inclusive at time of surgery.
3. Is willing and able to comply with the study plan and sign the Patient Informed Consent Form

Exclusion Criteria:

1. Has presence of active malignancy.
2. Has overt or active bacterial infection, either local or systemic.
3. Is mentally incompetent.
4. Is a prisoner.
5. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
6. Is pregnant or plan to be pregnant during the course of the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Hospitalization cost | 12 months
  Total medical costs including index surgery and re-admissions over 5 years

SECONDARY OUTCOMES:
Pain scales | 6, 12, 24, 36, 48 and 60 months
  Pain scales for back and leg pain (0 to 10)
Oswestry Low Back Pain Disability Questionnaire | 6, 12, 24, 36, 48 and 60 months
  Low back disability
Short Form 6D | 6, 12, 24, 36, 48 and 60 months
  Utility measure
EurQOL 5d | 6, 12, 24, 36, 48 and 60 months
  Utility measure
Readmissions | 90 days
  Number of readmissions 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Glassman, MD, Principal Investigator — Norton Leatherman Spine Center
Locations (1):
- Norton Leatherman Spine Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual level data.